CLINICAL TRIAL: NCT00861653
Title: Atherosclerotic Plaque Characterization Using Multispectral, Multicontrast High Resolution Cardiovascular Magnetic Resonance Imaging
Brief Title: Atherosclerotic Plaque Characterization
Acronym: APC
Status: Completed | Type: Observational
Sponsor: Piedmont Healthcare (Other)
Responsible Party: Sarah Rinehart, MD, Sarah Rinehart, MD
Other Study IDs: P06-31
Record Dates: First submitted 2009-03-11; First posted 2009-03-13 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis; Subjects diagnosed with atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and tissue samples are collected for markers of inflammation and gene chip analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to utilize high-resolution CMR carotid imaging for the characterization of carotid wall volumes and plaque content in patients with clinical significant carotid atherosclerosis. Patients who are scheduled to undergo an imaging procedure will be recruited from the cath lab. Upon enrollment, blood samples conventional and genetic profiling will be collected. For patients undergoing a carotid endarterectomy, tissue from the carotid vessel will be collected during their procedure. Comparison of the MR images with tissue and/or blood samples will be made. Length of time in the study will be approximately 1 day. There will be no study-related patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age range >17 years of age
* Surgical carotid artery disease
* Provide written informed consent and Authorization for Use/Disclosure of PHI

Exclusion Criteria:

* History of carotid trauma
* History of middle or large vessel vasculitis
* Refusal to provide written informed consent and Authorization for
* Use/Disclosure of PHI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with atherosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-10; Primary Completion 2011-08 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Characterization of plaque that is found in the carotid walls of patients who have atherosclerosis | 2 years post study initiation

SECONDARY OUTCOMES:
To evaluate the effectiveness of MR imaging in identifying these plaque characteristics | 2 Years Post Study Initiation

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rinehart, MD, Principal Investigator — Piedmont Healthcare
Locations (1):
- Piedmont Hospital, Atlanta, Georgia, United States